CLINICAL TRIAL: NCT07351799
Title: The Impact of Mindfulness and Meditation Based Lactation Education on Maternal Breastmilk in the Neonatal ICU: Intervention Study
Brief Title: Mindfulness and Meditation Based Lactation Education on Maternal Breastmilk in the Neonatal ICU
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ashley E. Thompson, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-013742
Record Dates: First submitted 2026-01-12; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Lactation; Mindfulness; NICU; Breastmilk; Neonatal; Meditation; Pumping, Breast; Cortisol; Oxytocin; Anxiety; Depression
Keywords: lactation; mindfulness; NICU; breastmilk; Neonatal; meditation; pumping, breast; cortisol; oxytocin; anxiety; Depression
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression; Anxiety Disorders; Depression | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): Mothers in the standard of care arm will undergo a standard lactation admission visit
  Interventions: Behavioral: Standard of Care
- Mindfulness-Based (Experimental): Mothers in the mindfulness-based arm will receive mindfulness-based lactation education along with a standard lactation admission visit
  Interventions: Behavioral: Mindfulness-based Intervention

INTERVENTIONS:
Behavioral: Standard of Care — No additional session with the lactation consultant will be provided beyond the standard of care lactation admission visit with a lactation consultant within 72 hours of their infant's admission to the NICU.
  On days 0, 10 and 20, participants will be asked to record pumping session times and breastmilk volumes expressed for 24 hours, collect salivary oxytocin sample and salivary cortisol sample at minute 4 of one pumping session, and fill out the GAD7, PSS, and PHQ-8 surveys.
  Arms: Standard of Care
Behavioral: Mindfulness-based Intervention — In addition to the standard of care lactation admission visit, participants will receive an additional session with the lactation consultant for mindfulness-based lactation education. Participants will also be provided with a pumping meditation audio recording that they will be asked to listen to at least once daily for the next 20 days.
  On days 0, 10 and 20, participants will be asked to record pumping session times and breastmilk volumes expressed for 24 hours, collect salivary oxytocin sample and salivary cortisol sample at minute 4 of one pumping session, and fill out the GAD7, PSS, and PHQ-8 surveys.
  In addition, the intervention group participants will also be asked to record the number of times they listened to the recording daily, minutes listened to recording daily, and time of day listened to recording.
  Arms: Mindfulness-Based

SUMMARY:
The purpose of this research is to investigate associations between mindfulness and meditation techniques and changes in maternal breastmilk in the mother pumping for her NICU infant.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > 20 years of age
* Read, write and understand English
* Infant NICU admit
* Infant birthplace of Rochester, MN (Mayo Clinic)
* Maternal adherence to pumping ≥ 8 times in 24 hours
* Mother enrolled within 72 hours of birth
* Gestational age of neonate at birth of < 34 0/7 weeks

Exclusion Criteria:

* Maternal extensive existing mindfulness practice
* Maternal breast/chest surgery
* Maternal polycystic ovarian syndrome (PCOS)
* Maternal current illicit substance abuse
* Diagnosis of maternal current severe mental health concerns
* Maternal multiple gestation (twins or higher order) pregnancy and delivery

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-11-02 (Estimated); Study Completion 2026-11-02 (Estimated)

PRIMARY OUTCOMES:
Change in breastmilk volume | Baseline, 10 days, 20 days
  Volume will be reported in milliliters (mL)

SECONDARY OUTCOMES:
Change in salivary oxytocin | Baseline, 10 days, 20 days
Change in salivary cortisol | Baseline, 10 days, 20 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Thompson, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials